CLINICAL TRIAL: NCT04133220
Title: Characterization of Endothelial Activation Hemostasis Disturbances and Severe Bleeding Events in Hyperleukocytic Acute Myeloid Leukemia
Brief Title: Endothelial Activation Hemostasis Disturbances and Severe Bleeding Events in Hyperleukocytic Acute Myeloid Leukemia
Acronym: HEAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 190002
Record Dates: First submitted 2019-07-01; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-06

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: hemostasis
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with acute myeloid leukemia, associated to hyper leukocytosis
- Control: Patients with acute myeloid leukemia, without hyper leukocytosis

SUMMARY:
Hyper-leukocytosis > 50.109/L is observed in 15% of acute myeloid leukemia (AML).

Level of hyper-leukocytosis is linearly associated with the incidence of life threatening complications that lead to the early death in 25% of these patients.

The HEAL project is a prospective, uni-centric, observational study that plans to include a cohort of 50 patients presenting de novo AML with hyper-leukocytosis (HL) (> 50.109/L) and 10 controls. The aim of the study is to describe the relative proportion of various hemostasis components disturbances, endothelium alterations, platelet dysfunction and to calculate cumulative incidence of hemorrhagic and thrombotic complications as well as overall survival of patients presenting with HL AML.

ELIGIBILITY:
Inclusion Criteria:

* De novo AML
* GB counts > 50 G/L
* Eligible for intensive chemotherapy
* no previous AML treatment

Exclusion Criteria:

* secondary AML
* relapse of AML
* Acute promyelocytic leukemia
* Previous antiplatelet or anticoagulant treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute myleoid leukemia associated to hyper-leukocytosis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of ICAM- | 12hours after chemotherapy initiation
  plasma concentration of ICAM-
Hemostasis / platelet and endothelial dysfunction parameter assessed by plasma concentration of Syndecan-1 | 12hours after chemotherapy initiation
  plasma concentration of Syndecan-1
Hemostasis / platelet and endothelial dysfunction parameter assessed by plasma concentration of vWF Ag | 12hours after chemotherapy initiation
  plasma concentration of vWF Ag
Hemostasis / platelet and endothelial dysfunction assessed by vWF activity | 12hours after chemotherapy initiation
  vWF activity
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of Fg | 12hours after chemotherapy initiation
  plasma concentration of Fg
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of t-PA | 12hours after chemotherapy initiation
  plasma concentration of t-PA
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of u-PA | 12hours after chemotherapy initiation
  plasma concentration of u-PA
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of e-Selectin | 12hours after chemotherapy initiation
  plasma concentration of e-Selectin
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of sCD40L | 12hours after chemotherapy initiation
  plasma concentration of sCD40L
Hemostasis / platelet and endothelial dysfunction parameter assessed by plasma concentration of IL6 | 12hours after chemotherapy initiation
  plasma concentration of IL6
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of AT | 12hours after chemotherapy initiation
  plasma concentration of AT
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of Fragments thrombin 1+2 | 12hours after chemotherapy initiation
  plasma concentration of Fragments thrombin 1+2
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of TAT complex | 12hours after chemotherapy initiation
  plasma concentration of TAT complex
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of plasmin-antiplasmin complex | 12hours after chemotherapy initiation
  plasma concentration of plasmin-antiplasmin complex
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of PAI-1 Ag | 12hours after chemotherapy initiation
  plasma concentration of PAI-1 Ag
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of PAI-1 activity | 12hours after chemotherapy initiation
  plasma concentration of PAI-1 activity
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of t-PA-PAI-1 complex | 12hours after chemotherapy initiation
  plasma concentration of t-PA-PAI-1 complex
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of ADAMTS13 Ag | 12hours after chemotherapy initiation
  plasma concentration of ADAMTS13 Ag
Hemostasis / platelet and endothelial dysfunction assessed by ADAMTS13 activity | 12hours after chemotherapy initiation
  ADAMTS13 activity
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of vWF:CB | 12hours after chemotherapy initiation
  plasma concentration of vWF:CB
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of Fibrin monomers | 12hours after chemotherapy initiation
  plasma concentration of Fibrin monomers
Hemostasis / platelet and endothelial dysfunction assessed by Prothrombine Time | 12hours after chemotherapy initiation
  Prothrombine Time
Hemostasis / platelet and endothelial dysfunction assessed by Activated Partial Thromboplastin Time [APTT] | 12hours after chemotherapy initiation
  Activated Partial Thromboplastin Time [APTT]
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of Factor IX | 12hours after chemotherapy initiation
  plasma concentration of Factor IX
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of Factor II | 12hours after chemotherapy initiation
  plasma concentration of Factor II
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of Factor VIII | 12hours after chemotherapy initiation
  plasma concentration of Factor VIII
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of Factor XII | 12hours after chemotherapy initiation
  plasma concentration of Factor XII
Hemostasis / platelet and endothelial dysfunction assessed by plasma concentration of Factor X | 12hours after chemotherapy initiation
  plasma concentration of Factor X

SECONDARY OUTCOMES:
Cumulative incidence of serious bleeding events | 1 month
  Time from inclusion to first serious bleeding event
Cumulative incidence of thrombotic events | 1 month
  Time from inclusion to first thrombotic event
Overall survival | 1 month
  Time from inclusion to death of any cause
ICU length of stay | 1 month
  duration of stay in ICU within the first month

IPD SHARING:
Plan to Share IPD: No